CLINICAL TRIAL: NCT00765375
Title: Double-Blind, Randomized, Placebo-Controlled Study to Determine the Safety and the Efficacy of Using Botulinum Neurotoxin Type A Injections for Subjects With Mild to Moderate Acne Vulgaris
Brief Title: Safety and Efficacy of the Use of Botox on Acne
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: DeNova Research (Other)
Responsible Party: Principal Investigator, Steven H. Dayan, Medical Director, DeNova Research
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BTX-D-001
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
Keywords: acne; Botox; cosmetic treatments
MeSH Terms: conditions — Acne Vulgaris | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botox and Placebo on each side of face (Experimental): Botulinum Neurotoxin Type A (Botox, 1.5-3 units/lesion); Bacteriostatic saline solution (0.11 cc/lesion)
  Interventions: Drug: Botulinum Neurotoxin Type A; Drug: Bacteriostatic saline

INTERVENTIONS:
Drug: Botulinum Neurotoxin Type A — 1.5-3 units of Botox/lesion
  Other Names: Botox
Drug: Bacteriostatic saline — .1 cc bacteriostatic saline/lesion

SUMMARY:
• To determine the safety and efficacy of Botox Treatment in subjects with mild to moderate acne vulgaris defined by the Investigator's Global Assessment (IGA)

DETAILED DESCRIPTION:
• 90 day trial, with botox being injected at baseline/screening visit. Photos will be taken throughout the study and patients will be evaluated by masked injector evaluator and a masked evaluator. Patient will complete a subject evaluation at each visit. Follow-up visits occur at Day 3, 7, 14, 30 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 and 50 years of age
* Not pregnant and negative pregnancy test, not planning on getting pregnant
* Mild to moderate bilateral acne lesions on the face
* Able to understand the requirements of the study and sign an Informed Consent Form
* Have the time and ability to complete the study and comply with instructions(i.e will be around for the duration of the study)
* Skin types I, II, III, IV and V

Exclusion Criteria:

* Subject has skin type VI
* Subject has a significant concurrent illness, such as diabetes, epilepsy, lupus or congestive heart disease
* Concurrent skin conditions affecting area to be treated
* Prior exposure to any serotype of botulinum toxin for any purpose in the 3 months immediately prior to study enrollment
* Prior surgery on the area to be treated within 3 months of initial treatment or during this clinical evaluation
* Open laceration, abrasion active cold sores or herpes sores, multiple dysplastic nevi in areas to be treated?
* Permanent or semi-permanent dermal filler treatment within the last 6 months
* Medium or deep depth chemical peel resurfacing procedure within 3 months of treatment or during this clinical evaluation
* Has used oral isotretinoin (Accutane) within 6 months, or use of topical isotretinoin within 3 months, of initial treatment or during this clinical evaluation
* Prior light /laser treatments at target locations within 3 months of enrollment or during the course of this clinical evaluation
* Any physical or mental condition which, in the investigator's opinion would make it unsafe for the subject to participate in the clinical evaluation
* Use of oral antibiotics for acne and/or medication that cause photosensitivity within 2 weeks of initial treatment
* Participation in a study of another investigational devices or drugs within 3 months of enrollment
* Subject shows symptoms of a hormonal disorder
* Subject cannot be treated for (past or present) any form of treatment of active cancer or having a history of skin cancer or any other cancer in the area to be treated
* Subject is currently using immunosuppressive medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD F.A.C.S., Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active on One Side, Placebo on the Other Side of Face: Botulinum Neurotoxin Type A (Botox) treatment on one side of the face and bacteriostatic saline solution (Placebo) on the other side of the face.
Period: Overall Study
Arm/Group | Active on One Side, Placebo on the Other Side of Face
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Active on One Side and Placebo on the Other Side of Face: Botulinum Neurotoxin Type A (Botox) on one side of face, and bacteriostatic saline solution on the other side of face.
Arm/Group | Active on One Side and Placebo on the Other Side of Face
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2.236)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Lesion Count From Baseline at 90 Days
Description: To determine the safety and efficacy of Botox Treatment in subjects with mild to moderate acne vulgaris defined by the Investigator's Global Assessment (IGA)
Time Frame: Baseline and 90 days
Population: All subjects completing Day 90 visit
Measure: Mean (Standard Deviation); unit: Lesions
Groups:
- 1- Active: Botulinum Neurotoxin Type A (Botox)
- 2- Placebo: Saline Solution
Arm/Group | 1- Active | 2- Placebo
Number analyzed (Participants) | 5 | 5
Lesions | 18.8 (7.33) | 15.8 (9.52)

ADVERSE EVENTS:
Arm/Group | 1- Active | 2- Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Study terminated after 5 subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes